CLINICAL TRIAL: NCT04301271
Title: Simvastatin add-on to Escitalopram in Patients With Comorbid Obesity and Major Depression: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Simvastatin add-on Treatment to Standard Antidepressant Therapy in Patients With Comorbid Obesity and Major Depression
Acronym: SIMCODE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other); University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christian Otte, Professor of Psychiatry, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIMCODE
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Depressive Disorder, Major; Obesity
MeSH Terms: conditions — Depressive Disorder, Major; Obesity | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin (Experimental): Simvastatin and Escitalopram
  Interventions: Drug: Simvastatin 40mg
- Placebo (Placebo Comparator): Placebo and Escitalopram
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Simvastatin 40mg — 12 weeks 40 mg Simvastatin add-on
  Other Names: Zocor; C10AA01
  Arms: Simvastatin
Drug: Placebo oral tablet — 12 weeks Placebo add-on
  Arms: Placebo

SUMMARY:
Major depressive disorder (MDD) and obesity are major contributors to impaired health worldwide. Statins are among the most prescribed medications with well-established safety and efficacy. Statins are recommended in primary prevention of cardiovascular disease, which has been linked to both MDD and obesity. Moreover, statins are promising candidates to treat MDD because a meta-analysis of pilot randomized controlled trials has found antidepressive effects of statins as adjunct therapy to antidepressants. However, no study so far has tested the antidepressive potential of statins in patients with MDD and comorbid obesity. Therefore, we hypothesize that Simvastatin add-on to standard antidepressant Escitalopram will improve depression to a greater extent than add-on placebo in patients with comorbid obesity and major depression. We will randomize 160 obese MDD patients at 8 recruiting centers to either Simvastatin or placebo as add-on to Escitalopram for 12 weeks. If successful, our trial would have immediate impact on clinical practice given the fact that Simvastatin and Escitalopram are available as inexpensive generic drugs with established safety.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is present
* The patient has the capacity to give consent (He/she is able to understand the nature and anticipated effects/side effects of the proposed medical intervention)
* The patient has a major depressive episode according to DSM 5 (Diagnostic and Statistical Manual of Mental Disorders 5th Edition)
* The patient has a score of ≥ 18 in the Montgomery-Asberg Depression Rating Scale (MADRS)
* The patient has a body mass index ≥ 30
* The patient's age is between 18 and 65 years (≥ 18 und ≤ 65)
* The patient has not given childbirth within the 6 months prior to study entry and is not breastfeeding
* In case of non-psychotropic medication: The patient received stable pharmacological medication for at least 14 days prior to study entry (any changes in medication dose or frequency of therapy must be answered with no)
* The patient did not take antidepressants during the last 7 days prior to study entry (discontinuation of effective medication to enable study participation is prohibited)
* The patient did not receive prior treatment with Escitalopram in index episode
* The patient had less than three (<3) trials with antidepressants in index episode
* The patient does not have a history of non-response to Escitalopram
* The patient did not receive treatment with ketamine, irreversible MAO inhibitor (e.g. tranylcypromine), electroconvulsive therapy (ECT) or other stimulatory treatments in index episode
* The patient does not meet any of the following criteria: schizophrenia, schizoaffective disorder, bipolar disorder
* The patient is not diagnosed with dementia and does not have moderate or severe impairment of general cognitive function according to clinical impression
* The patient does not have clinically relevant elevated liver enzymes [GOT or GPT > 3 x upper limit normal (ULN)] and does not have elevated Carbohydrate Deficient Transferrin (CDT) ≥ 2.4 %
* The patient does not meet the criteria for alcohol use disorder (DSM-5: 303.90; ICD-10: F10.20) or substance use disorder (DSM-5: 304; ICD-10: F11.20 - F19.20) in M.I.N.I. for DSM-5 and a urine/serum drug screening is negative (except for benzodiazepines and opiates)
* The patient does not have a history of suicide attempt
* The patient does not have diagnosed epilepsy or increased bleeding diathesis or a history of angle closure glaucoma or other glaucomas
* The patient did not have bariatric surgery prior to study entry
* The patient does not have a known allergy or contraindication against Escitalopram or Simvastatin
* The patient does not meet any of the following criteria: hereditary muscle disease, known history of rhabdomyolysis, elevated creatine kinase (CK) outside of the sex-specific reference intervals, history of muscular symptoms under treatment with statins or fibrates
* The patient does not have elevated TSH level outside of the age- and sex-specific refer-ence intervals.
* The patient does not have insulin-dependent diabetes mellitus
* The patient does not have uncontrolled hepatic disorder, renal or cardiovascular disease
* The patient does not have untreated hypothyroidism
* The patient does not have a history of myocardial infarction or stroke
* The patient does not have symptomatic peripheral arterial disease
* The patient does not have monogenic familial hypercholesterolemia
* The patient does not have clinically significant laboratory abnormalities
* The patient did not participate in other interventional trials during the 6 months before and at the time of this trial
* The patient is not an employee of the investigator study site, or a family member of the employees or the investigator, or otherwise dependent on the sponsor, the investigator or the investigator study site

Exclusion Criteria:

* The patient has current use of statins (for visits 2-6 applies: except for IMP Simvastatin)
* The patient has current use of antidepressants (for visits 2-6 applies: except for standard medication Escitalopram)
* The patient has acute suicidal tendencies (MADRS Item 10 > 4)
* The patient uses potent CYP3A4-inhibitors (e.g. clarithromycin, erythromycin, HIV protease inhibitors - see "Risks, adverse drug reactions, drug interactions, restrictions, contraindications, procedures in case of emergency")
* The patient uses potent CYP3A4 inductors (Carbamazepine, Efavirenz, Nevirapine, Etravirine).
* The patient uses Fibrates, Amiodarone, Amlodipine, Verapamil, Fluconazol, Diltiazem, Fusidic acid, Niacin or Lomitapide or BCRP-Inhibitors (e.g. Elbasvir or Grazoprevir)
* The patient uses Gemfibrozil, Ciclosporin or Danazol
* The patient has known hypersensitivity to other ingredients of Simvastatin and Escitalopram [butylated hydroxyanisole, microcrystalline celluose, citric acid, starch, lactose, magnesium stearate, hypromellose, talc, titanium dioxide, iron oxides, colloidal silicon dioxide, croscarmellose sodium, polyethylene glycol]
* The patient uses medication that is associated with QTc-prolongation [antiarrhythmics class IA and III, antipsychotics (e.g. Haloperidol), phenothiazines, tricyclic antidepressants, antibiotics (e.g. Moxifloxacin), and certain antihistaminergic drugs (e.g. Astemizol, Mizolastine)]
* The patient has clinically significant abnormalities in 12-lead ECG (e.g. QTc-prolongation ≥ 500 ms or increase ≥ 60 ms from baseline visit)
* The patient is pregnant
* The patient with childbearing potential is not willing to use an acceptable form of contraception (defined as Pearl index < 1)
* The patient has current use of psychotropic medication (e.g. antipsychotics, anticonvulsants, lithium or St. John's Wort) except for benzodiazepines, non-benzodiazepines and opiates
* The patient uses nonselective, irreversible monoamine oxidase (MAO) inhibitor (e.g. Tranylcypromine) or selective, reversible inhibitor of monoamine oxidase A (e.g. Moclobemide) or the nonselective, reversible monoamine oxidase inhibitor Linezolid
* The patient is unwilling to consent to saving, processing and propagation of pseudonymized medical data for study reasons
* The patient is legally detained in an official institution

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Change score in MADRS (Montgomery-Asberg-Depression Rating Scale) | 12 weeks
  The MADRS is a rating scale to measure depression severity. Each MADRS item is rated on a 0 to 6 scale. Total score range from 0-60, where higher MADRS scores indicate higher levels of depressive symptoms.

SECONDARY OUTCOMES:
MADRS-response | 12 weeks
  Response is defined as 50% MADRS score reduction at week 12 from baseline.
MADRS-remission | 12 weeks
  Remission is defined as a MADRS score less than 10 at week 12.
MADRS-MCID | 12 weeks
  MADRS Minimal Clinically Important Difference represents the smallest improvement that is considered meaningful by the patient. Empirically, the MCID using the MADRS has been identified as a change from baseline between 1.6 - 1.9 at week 12.
Change score in BDI-II (Beck Depression Inventory-II) | 12 weeks
  The Beck Depression Inventory-II (BDI-II) is a 21-item validated instrument for the self-report of depressive symptoms, with individual item scores summed to yield a total possible BDI score that ranges from 0-63. BDI scores from 0-13 suggest absent to minimal depressive symptoms, from 14-19 mild symptoms, from 20-28 moderate symptoms, and from 29-63 severe symptoms.
BDI-II-MCID | 12 weeks
  BDI-II Minimal Clinically Important Difference represents the smallest improvement that is considered meaningful by the patient.
Change score in PGIC (Patients' Global Impression of Change Scale) | 12 weeks
  Participant rated instrument to measure participant's change in overall status on a scale of 0 to 7; range from 1 (very much improved) to 7 (very much worse).
Change score in CGI-S (Clinicians' Global Impression of Severity of Illness) | 12 weeks
  The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. The CGI-S permits a global evaluation of the participant's condition at a given time.
CGI-I (Clinicians' Global Impression of Improvement ) | 12 weeks
  Clinician rated instrument to measure clinicians' change in overall status on a scale of 0 to 7; range from 1 (very much improved) to 7 (very much worse).
EQ-5D-3L (EuroQol-5 Dimensions-3 Levels Questionnaire) | 12 weeks
  Generic instrument of quality of life related to health. It contains five dimensions of health (mobility, personal care, daily activities, pain / discomfort and anxiety / depression) and each of them has three levels of seriousness (without problems, some problems or moderate problems and serious problems).
  The second part of the EQ-5D is a Visual Analogue Scale (VAS) of 20 centimeters, millimeter, ranging from 0 (worse health status imaginable) to 100 (best imaginable health status). In it, the individual must mark the point in the vertical line that best reflects the assessment of their global health status today.
SOFAS (Social and Occupational Functioning Assessment Scale) | 12 weeks
  The SOFAS is a rating scale used to determine social functioning; range from 0-100. A higher score represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Otte, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (9):
- Germany (9):
  - Charité - Universitätsmedizin Berlin, Klinik für Psychiatrie und Psychotherapie, Berlin
  - Charité - Universitätsmedizin Berlin, Medizinische Klinik mit Schwerpunkt Psychosomatik, Berlin
  - Universitätsklinikum Frankfurt, Klinik für Psychiatrie, Psychosomatik und Psychotherapie, Frankfurt
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Psychiatrie, Sozialpsychiatrie und Psychotherapie, Hanover
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Psychiatrie und Psychotherapie, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Zentrum für Integrative Psychiatrie - Klinik für Psychiatrie und Psychotherapie, Lübeck
  - Helios Hanseklinikum Stralsund Klinik und Poliklinik für Psychiatrie, Psychotherapie und Psychosomatik, Stralsund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otte C, Chae WR, Dogan DY, Piber D, Roepke S, Cho AB, Trumm S, Kaczmarczyk M, Brasanac J, Wingenfeld K, Koglin S, Wieditz J, Junghanns K, Lucht M, Prvulovic D, Kruger THC, Terock J, Haaf M, Hofmann T, Mauche N, Klein JP, Grabe HJ, Reif A, Kahl KG, Janowitz D, Leicht G, Hinkelmann K, Strauss M, Friede T, Gold SM. Simvastatin as Add-On Treatment to Escitalopram in Patients With Major Depression and Obesity: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Aug 1;82(8):759-767. doi: 10.1001/jamapsychiatry.2025.0801. PMID 40465256
- [Derived] Otte C, Chae WR, Nowacki J, Kaczmarczyk M, Piber D, Roepke S, Marschenz S, Lischewski S, Schmidt S, Ettrich B, Grabe HJ, Hegerl U, Hinkelmann K, Hofmann T, Janowitz D, Junghanns K, Kahl KG, Klein JP, Krueger THC, Leicht G, Prvulovic D, Reif A, Schoettle D, Strauss M, Westermair A, Friede T, Gold SM. Simvastatin add-on to escitalopram in patients with comorbid obesity and major depression (SIMCODE): study protocol of a multicentre, randomised, double-blind, placebo-controlled trial. BMJ Open. 2020 Dec 1;10(12):e040119. doi: 10.1136/bmjopen-2020-040119. PMID 33262189

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT04301271/Prot_SAP_000.pdf